CLINICAL TRIAL: NCT02159638
Title: Accuracy of Two CGM Systems Tested Simultaneously in Ambulatory Patients With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vastra Gotaland Region (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGFOUREG-387191
Record Dates: First submitted 2014-06-05; First posted 2014-06-10 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2014-06

CONDITIONS: Diabetes Mellitus, Type 1; Blood Glucose
Keywords: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Insulin-Dependent; Endocrine System Diseases; Blood glucose; Blood Glucose, Self-Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus; Endocrine System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- comparisson CGM accuracy (Other): Each patient will have both subcutaneous tissue CGM sensors (Guardian Enlite sensor and Dexcom G4 Platinum sensor) inserted at the same time. The HemoCue Analyser- venous blood and finger-stick blood in cuvette, will be used to measure the concentration of glucose
  Interventions: Device: Guardian Enlite sensor; Device: Dexcom G4 platinum sensor

INTERVENTIONS:
Device: Guardian Enlite sensor — Sensor insertion
Device: Dexcom G4 platinum sensor — Sensor insertion

SUMMARY:
Continuous glucose monitoring (CGM) is a tool used in the treatment of patients with type 1 diabetes. A continuous glucose monitor (CGM) is a subcutaneous tissue sensor, which provides a tissue fluid glucose measurement every 1 to 5 minutes. Since CGM measure the glucose level by a sensor in subcutaneous tissue, there is uncertainty in the estimation of blood glucose levels. The accuracy of a certain CGM system can be assessed by comparing the glucose levels estimated by CGM with measured glucose levels in plasma. In the current study, we will compare the accuracy of the 2 CGM systems available on the market for clinical use in patients with type 1 diabetes. The aim of the current study is to evaluate effectiveness, safety and treatment satisfaction with 2 different CGM systems among adult type 1 diabetic patients.

DETAILED DESCRIPTION:
Each study patient will have both subcutaneous tissue CGM sensors inserted. Each sensor will produce a maximum of 1,440 tissue fluid glucose measurements per 24 hours and 8,460 measurements during the 6 days in study. The plan is to study 36 to 50 ambulatory patients during the hole study period. The two CGM data sets (DexCom4G and Medtronic Enlite) will be compared to each other and the time-matched reference blood glucose measurements.

The HemoCue Analyser- venous blood and finger-stick blood in cuvette, will be used to measure the concentration of glucose.

Each ambulatory patient will sample capillary blood and measure the concentration of glucose 6 to 10 times per day for max 6 days. The concentration of finger-stick capillary blood glucose will be measured using the HemoCue meter in their daily living and additionally a HemoCue Analyser at research visits using a lancet. Each patient will be admitted to the clinical research unit (CRU) for 7 measurements of venous samples at two occasions: on day 1-3 and 4-6 of the study with an interval of at least 15 minutes. An intravenous catheter will be inserted to facilitate blood sample acquisition each of these days of study. Three capillary finger-stick blood will be sampled at these 2 occasions, 1 at the first venous measurement (one day of days 1-3) and one at the last venous sample (one day of days 4-6).

Blood sample acquisition and handling will be standardized to minimize pre-analytical error.

The sensor insertion sites will be observed to detect bleeding, inflammation and infection of the skin or subcutaneous tissue. Insertion sites will be photographed if any abnormal findings exist at the end of the study for the individual patient.

The subjects will record self monitoring of blood glucose (SMBG), meal, and activity data in a written diary.

ELIGIBILITY:
Inclusion Criteria:

1. Type 1 diabetes
2. Adult patients, age 18 or older and <75 years.
3. Written Informed Consent

Exclusion Criteria:

1. Pregnancy
2. Patients with severe cognitive dysfunction or other disease which makes CGM use difficult.
3. Patients requiring continuous use of paracetamol. Paracetamol must not have been used

   the week before the study and shall not be used during the duration because it disturbs the

   interpretation of blood glucose levels estimated by the DexCom4G. However, other pain

   killers can be used throughout the study period.
4. Current CGM use
5. History of allergic reaction to any of the CGMS materials

   or adhesives in contact with the skin.
6. History of allergic reaction to chlorhexidine or alcohol

   anti-septic solution.
7. Abnormal skin at the anticipated glucose sensor

attachment sites (excessive hair, burn, inflammation,

infection, rash, and/or tattoo).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2013-05; Primary Completion 2014-07-01 (Actual); Study Completion 2014-09-01 (Actual)

PRIMARY OUTCOMES:
Difference between the two CGM systems compared to capillary glucose value | 6 days
  Primary efficacy analysis will be investigating whether there is a statistically significant difference between the two CGM systems with respect to mean absolute relative difference (MARD) of estimated capillary glucose value over the whole study period.

SECONDARY OUTCOMES:
the accuracy of the 2 CGM systems during each studied time interval (day 1-3 and day 4-6) | day 1-3 and day 4-6
  Accuracy of all estimated capillary glucose values (registered both during days 1-3 and days 4-6) of DexCom 4G system (DexCom sensor) vs Guardian Real-Time system (Enlite sensor) system compared to the capillary reference blood glucose measured with HemoCue.
the accuracy of the 2 CGM systems for hypoglycaemia | 6 days
  Accuracy in estimating capillary glucose levels <4 registered both during days 1-3 and days 4-6 of DexCom 4G system (DexCom sensor) vs Guardian Real-Time system (Enlite sensor) system compared to the capillary reference blood glucose measured with HemoCue(hypo, normoglycaemia and hyperglycaemia)
the accuracy of the 2 CGM systems for normoglycaemia | 6 days
  Accuracy in estimating capillary glucose levels of 4.0-10.0 mmol/l registered both during days 1-3 and days 4-6 of DexCom 4G system (DexCom sensor) vs Guardian Real-Time system (Enlite sensor) system compared to the capillary reference blood glucose measured with HemoCue
the accuracy of the 2 CGM systems for hyperglycaemia | 6 days
  Accuracy in estimating capillary glucose levels >14.0 mmol/l registered both during days 1-3 and days 4-6 of DexCom 4G system (DexCom sensor) vs Guardian Real-Time system (Enlite sensor) system compared to the capillary reference blood glucose measured with HemoCue
Evaluation of two CGM systems from questionnaire | day 6
  Evaluation of DexCom 4G system (DexCom sensor) vs Guardian Real-Time system (Enlite sensor) from questionnaire

CONTACTS AND LOCATIONS:
Locations (2):
- Sweden (2):
  - NU-hospital Organisation, Trollhättan
  - Uddevalla hospital, Uddevalla

REFERENCES:
- [Derived] Matuleviciene V, Joseph JI, Andelin M, Hirsch IB, Attvall S, Pivodic A, Dahlqvist S, Klonoff D, Haraldsson B, Lind M. A clinical trial of the accuracy and treatment experience of the Dexcom G4 sensor (Dexcom G4 system) and Enlite sensor (guardian REAL-time system) tested simultaneously in ambulatory patients with type 1 diabetes. Diabetes Technol Ther. 2014 Nov;16(11):759-67. doi: 10.1089/dia.2014.0238. Epub 2014 Sep 18. PMID 25233297